CLINICAL TRIAL: NCT06061445
Title: A Study to Evaluate the Effects of Radiotherapy Combined With Tyrosine Kinase Inhibitor (TKI) and Anti-PD-1 Antibody for Stage IIIA Hepatocellular Carcinoma With Portal Vein Tumor Thrombus(PVTT)
Brief Title: Radiotherapy Combined With TKI and Anti-PD-1 Antibody for Stage IIIA Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTI
Record Dates: First submitted 2023-08-14; First posted 2023-09-29 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-07

CONDITIONS: Stage IIIA Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Radiotherapy Combined with TKI and Anti-PD-1 Antibody
  Interventions: Combination Product: Radiotherapy combined with TKI and Anti-PD-1 Antibody

INTERVENTIONS:
Combination Product: Radiotherapy combined with TKI and Anti-PD-1 Antibody — After signing informed consent, patients received Anti-PD-1 Antibody 200 mg intravenously on the first day of each cycle, Q3W; Tyrosine Kinase Inhibitor (TKI) was administration started on the first and continually administered until disease progression developed or serious treatment-related toxicity occurred; Cancer thrombus radiotherapy treatment: For the portal vein cancer thrombus site (Total dose 25-30Gy, times 5-6) , Treatment usually starts within 7 days and ends within 1 week after the first cycle of injection of anti PD-1 inhibitors.

SUMMARY:
The purpose of this clinical research study is to investigate the efficacy and safety of Radiotherapy Combined with TKI and Anti-PD-1 Antibody for Stage IIIA Hepatocellular Carcinoma with Portal Vein Tumor Thrombus(PVTT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hepatocellular carcinoma who strictly meet the clinical diagnostic criteria of the "Guidelines for the Diagnosis and Treatment of Primary Liver Cancer" (2022 edition) or who have been confirmed by histopathology or human cytology, There was at least one measurable lesion (spiral CT scan length ≥10mm or malignant lymph node short diameter ≥15mm according to RECIST1.1 standard);
* Patients with advanced primary hepatocellular carcinoma who have not received systematic treatment and cannot be surgically resectable;
* CNLC was divided into stage IIIA, VP1-3 type;
* Child-Pugh classification of liver function is grade A (5-6 points);
* ECOG PS score 0-1;
* Expected survival ≥12 weeks;
* Patients with active hepatitis B virus (HBV) infection must be willing to receive antiviral treatment throughout the study period; Hepatitis C virus (HCV) ribonucleic acid (RNA) positive patients must receive antiviral therapy according to standard local treatment guidelines and have liver function within CTCAE level 1 elevation;
* The major organs function normally and meet the following criteria :

  1. The blood routine examination criteria should meet :(no blood transfusion within 14 days)

     1. Hemoglobin (HB)≥90g/L,
     2. White blood cell count (WBC)≥3×109/L,
     3. Absolute neutrophil count (ANC)≥1.5×109/L,
     4. platelets (PLT)≥75×109/L;
  2. Biochemical examination should meet the following criteria:

  <!-- -->

  1. Bilirubin (BIL)< 1.5 times the upper limit of normal value (ULN);
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase AST<5ULN;
  3. Serum creatinine (Cr)≤1.5ULN
* Women of childbearing age must have a negative pregnancy test (serum) or urine HCG test within 7 days prior to admission and be willing to use an appropriate method of contraception during the trial and 8 weeks after the last dose of the test drug; For males, they should be surgically sterilized or agree to use appropriate methods to avoid pregnancy during the trial and for 8 weeks after the last dose of the trial drug;
* The subjects voluntarily joined the study, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Pregnant or lactating women;
* Patients with autoimmune diseases, organ/hematopoietic stem cell transplantation, or other malignancies (except cured cutaneous basal cell carcinoma and cervical carcinoma in situ);
* Patients with consciousness disorder or inability to cooperate with treatment, combined with mental illness;
* Patients with a history of epigastric radiotherapy;
* Patients who fail to follow dose limits for vital organs in the radiotherapy program, including patients with normal liver tissue less than 700 ml in the radiotherapy program;
* Patients who have participated in other clinical trials in the past three months;
* Previously received targeted therapy or other PD-1/PD-L1 inhibitor therapy;
* Received major surgery or chemotherapy, radiation therapy or other focal systemic therapy within 1 month before enrollment;
* Immunosuppressive agents or systemic hormone therapy (dose >10mg/ day prednisone or other therapeutic hormones) were used within 14 days before enrollment to achieve immunosuppression;
* Liver function was classified as Child-Pugh C, which could not be improved by liver protection treatment.
* Esophageal (fundus) varices rupture and bleeding within 1 month before treatment.
* Uncorrectable coagulation dysfunction and severe blood abnormalities, with a tendency to severe bleeding. Platelet count <50×109/L and severe coagulation dysfunction can not withstand surgery (anticoagulant therapy and/or anticoagulant drug use should be stopped more than 1 week before radiotherapy);
* Refractory ascites, bad fluid;
* Active infection, especially inflammation of the biliary system;
* Severe liver, kidney, heart, lung, brain and other major organ failure;
* People who have been allergic to any component of PD-1 monoclonal antibody or other similar experimental drugs;
* Have high blood pressure and can not be reduced to normal by antihypertensive medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | the date of first administration to the subject's death from various causes
  Overall survival (OS) was measured from the initiation of transarterial therapy to the date of death or the last follow-up.
ORR | The best efficacy recorded between the date of first administration and the date of objective recording of progress according to mRECIST 1.1 criteria or the date of initiation of subsequent antitumor therapy, whichever occurs first
  Assessed according to the modified Response Evaluation Criteria in Solid Tumors Version 1.1, undergoing enhanced CT/MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China